CLINICAL TRIAL: NCT00603720
Title: PET Detection of the Effects of Aging on the Human Heart. Aim#1-Impact of Aging on Myocardial Remodeling: Role of Nitric Oxide
Brief Title: Role of Nitric Oxide in the Impact of Aging on Myocardial Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AG0086; 5R01AG015466-08 (NIH); 05-0810 (Registry Identifier: HRPO); RDRC# 482F (Other: RDRC); GCRC# 1002 (Other: GCRC)
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Diseases
Keywords: PET; Heart metabolism; Nitric oxide; Myocardial remodeling
MeSH Terms: conditions — Cardiovascular Diseases | interventions — NG-Nitroarginine Methyl Ester; Arginine; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- L-Name in Young (Active Comparator): 20 individuals age 18-35 will be getting an infusion of L-NAME (a nitric oxide inhibitor) during 3 separate PET study days, then a 10-minute infusion of L-arginine to reverse effects of L-NAME.
  Interventions: Drug: L-NAME
- Phenylephrine (Active Comparator): 25 individuals age 18-35 will be getting an infusion of phenylephrine (primarily an alpha agonist) during 3 separate PET study days
  Interventions: Drug: Phenylephrine
- L-arginine in Young (Active Comparator): 20 individuals age 18-35 will be getting an infusion of L-arginine 125 mcg/kg/min for 120 to 140 minutes during 3 separate PET study days
  Interventions: Drug: L-Arginine
- L-arginine in Old (Active Comparator): 20 individuals age 60-75 will be getting an infusion of L-arginine 125 mcg/kg/min for 120 to 140 minutes during 3 separate PET study days
  Interventions: Drug: L-Arginine
- L-NAME in Old (Experimental): 20 individuals age 60-75 will be getting an infusion of L-NAME (a nitric oxide inhibitor) during 3 separate PET study days, then a 10-minute infusion of L-arginine to reverse effects of L-NAME
  Interventions: Drug: L-NAME

INTERVENTIONS:
Drug: L-NAME — nitric oxide synthase inhibitor 4mg/kg infusion over 30-60 minutes prior to PET imaging
  Other Names: N (G)-nitro-L- arginine methyl ester
  Arms: L-NAME in Old; L-Name in Young
Drug: L-Arginine — aids in nitric oxide production
  Other Names: 2-Amino-5-guanidinopentanoic acid
  Arms: L-arginine in Old; L-arginine in Young
Drug: Phenylephrine — alpha agonist; 10 μg/kg/min infusion during PET study
  Other Names: (R)-3-[-1-hydroxy-2-(methylamino)ethyl]phenol
  Arms: Phenylephrine

SUMMARY:
The purpose of this study is to determine, with Positron Emission Tomography (PET), the role of nitric oxide in the age-associated effect on fatty acid and glucose delivery on myocardial substrate metabolism.

DETAILED DESCRIPTION:
Aging is associated with an increased incidence and severity of various cardiovascular disorders. Previously, our laboratory has demonstrated an age-related shift in the substrates used by the heart for metabolism from primarily fatty acids to primarily glucose. Furthermore, other institutions have demonstrated that a similar shift can be induced, in animal models, with specific nitric oxide synthase inhibitors, such as L-NAME (N-Nitro-L-Arginine Methyl Ester). Our hypothesis is that a reduction in nitric oxide (NO) synthesis is responsible for the age-related shift in heart function. Accordingly, we aim to demonstrate, in young patients, an acute, transient shift in substrate use from fatty acids to glucose with L-NMMA (citrate) in association with depressed heart function. Also, we aim to demonstrate in the elderly an acute, transient shift in substrate use from glucose to fatty acids with L-arginine, in association with improved cardiac function. These results will demonstrate a portion of the mechanism for the age-related shift in substrate utilization.

Each participant will undergo a screening visit which will include a Glucose Tolerance Test, an echocardiogram in conjunction with a treadmill stress test to exclude cardiac disease, and baseline blood work. Then each patient will have 3 PET study days, each lasting about 5-6 hours. During this time, the patient will have two IVs (one in each arm). They will have 4 injections of different radioactive isotopes (015 Water, C11 Acetate, C11 Glucose, and C11 Palmitate). After each injection, about 8-10 blood samples will be drawn over the course of about ½ to 1 hour of time. In between each injection, there will be about an hour break for the patient to rest and move around. During one of the breaks, the patient will have another echocardiogram. On the day 2 and 3 PET, the patient will have a 30-60 minute infusion of L-NAME. Then the PET study will commence. After the study is over the participant will have a 10-minute infusion of L-arginine to reverse the effects of L-NAME.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35 or 60-75
* Normal glucose tolerance test
* Normal plasma fasting lipid panel (fasting total cholesterol less than 220 mg/dL)
* Normal rest/stress echocardiogram
* BMI (Body Mass Index) less than 30 kg/m2

Exclusion Criteria:

* Coronary artery disease
* High blood pressure
* Current smoker
* Diabetes mellitus
* Cardiovascular disease (signs and symptoms of any kind)
* History of stroke, peripheral vascular disease, or arrhythmia
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogawa T, Spina RJ, Martin WH 3rd, Kohrt WM, Schechtman KB, Holloszy JO, Ehsani AA. Effects of aging, sex, and physical training on cardiovascular responses to exercise. Circulation. 1992 Aug;86(2):494-503. doi: 10.1161/01.cir.86.2.494. PMID 1638717
- [Background] Olivetti G, Melissari M, Capasso JM, Anversa P. Cardiomyopathy of the aging human heart. Myocyte loss and reactive cellular hypertrophy. Circ Res. 1991 Jun;68(6):1560-8. doi: 10.1161/01.res.68.6.1560. PMID 2036710
- [Background] Coughlin SS, Neaton JD, Sengupta A, Kuller LH. Predictors of mortality from idiopathic dilated cardiomyopathy in 356,222 men screened for the Multiple Risk Factor Intervention Trial. Am J Epidemiol. 1994 Jan 15;139(2):166-72. doi: 10.1093/oxfordjournals.aje.a116978. PMID 8296783
- [Background] Haldeman GA, Croft JB, Giles WH, Rashidee A. Hospitalization of patients with heart failure: National Hospital Discharge Survey, 1985 to 1995. Am Heart J. 1999 Feb;137(2):352-60. doi: 10.1053/hj.1999.v137.95495. PMID 9924171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | L-Name in Young | Phenylephrine | L-arginine in Young | L-arginine in Old | L-NAME in Old
Started | 10 | 10 | 12 | 10 | 12
Completed | 10 | 10 | 12 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-Name in Young | Phenylephrine | L-arginine in Young | L-arginine in Old | L-NAME in Old | Total
Number analyzed (Participants) | 10 | 10 | 12 | 10 | 12 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 12 | 10 | 12 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 12 | 10 | 12 | 54
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 12 | 10 | 12 | 54

OUTCOME MEASURES:

1. Primary Outcome: Effect of NO Inhibition on Myocardial Substrate Metabolism in Humans
Description: Determine in young healthy volunteers the extent to which acute inhibition of nitric oxide production will effect a shift in myocardial substrate utilization characterized as a decline in myocardial fatty acid oxidation, and perhaps myocardial fatty acid utilization, and increase in myocardial glucose uptake, and whether these changes are associated with a decline in LV function.
Time Frame: 1-3 months
Population: PI left institution. Efforts were made to access the data, without success so there is no access to the data.
Measure: Mean (90% Confidence Interval); unit: percentage of substrate
Arm/Group | L-Name in Young | Phenylephrine | L-arginine in Young | L-arginine in Old | L-NAME in Old
Number analyzed (Participants) | 10 | 10 | 12 | 10 | 12
percentage of substrate | NA [NA to NA] — PI left institution. There is no access to the data. | NA [NA to NA] — PI left institution. There is no access to the data. | NA [NA to NA] — PI left institution. There is no access to the data. | NA [NA to NA] — PI left institution. There is no access to the data. | NA [NA to NA] — PI left institution. There is no access to the data.

ADVERSE EVENTS:
Time Frame: 1 to 3 months
Groups:
- L-Name in Young: 10 individuals age 18-35 will be getting an infusion of L-NAME (a nitric oxide inhibitor) during 3 separate PET study days, then a 10-minute infusion of L-arginine to reverse effects of L-NAME.
  L-NAME: nitric oxide synthase inhibitor 4mg/kg infusion over 30-60 minutes prior to PET imaging
- Phenylephrine: 10 individuals age 18-35 will be getting an infusion of phenylephrine (primarily an alpha agonist) during 3 separate PET study days
  Phenylephrine: alpha agonist; 10 μg/kg/min infusion during PET study
- L-arginine in Young: 12 individuals age 18-35 will be getting an infusion of L-arginine 125 mcg/kg/min for 120 to 140 minutes during 3 separate PET study days
  L-Arginine: aids in nitric oxide production
- L-arginine in Old: 12 individuals age 60-75 will be getting an infusion of L-arginine 125 mcg/kg/min for 120 to 140 minutes during 3 separate PET study days
  L-Arginine: aids in nitric oxide production
- L-NAME in Old: 10 individuals age 60-75 will be getting an infusion of L-NAME (a nitric oxide inhibitor) during 3 separate PET study days, then a 10-minute infusion of L-arginine to reverse effects of L-NAME
  L-NAME: nitric oxide synthase inhibitor 4mg/kg infusion over 30-60 minutes prior to PET imaging
Arm/Group | L-Name in Young | Phenylephrine | L-arginine in Young | L-arginine in Old | L-NAME in Old
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/12 | 0/10 | 0/12

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes